CLINICAL TRIAL: NCT04915794
Title: The Effects of Simulation on Knowledge and Self-efficacy of Nurses and Midwives in Preeclamptic Pregnancy Care Education
Brief Title: Preeclamptic Pregnancy Care Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gözde Küğcümen, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10377247
Record Dates: First submitted 2021-01-26; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Preeclampsia; Nurse's Role
Keywords: Preeclampsia; Self-efficacy
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation based education (Experimental): Simulation is a technique that creates a situation or environment that allows people to experience the representation of a real event, practice, learn, evaluate, test, or gain an understanding of systems or human actions
  Interventions: Other: Simulation of preeclamptic pregnancy care
- Traditional education (No Intervention): Necessary procedures explained theoretically

INTERVENTIONS:
Other: Simulation of preeclamptic pregnancy care — It is an important step in providing safe care to patients, as a learning environment is provided in which environmental risks are minimized with simulation applications. Simulation-based trainings are environments that allow each student to learn, equitable, based on adult learning principles, and open to different learning styles. In these environments, interests and needs are defined together by the learner and the educator. By keeping the experiences of the learner at the forefront, the opportunity is given to learn by doing and is supported with feedback.
  Arms: Simulation based education

SUMMARY:
The aim of this study is to evaluate the effect of simulation training in nurses and midwives on knowledge and self-efficacy regarding preeclamptic pregnancy care.

It is an important step in providing safe care to patients, as a learning environment is provided in which environmental risks are minimized with simulation applications. Simulation-based trainings are environments that allow each student to learn, equitable, based on adult learning principles, and open to different learning styles. The interests and needs in these environments are defined together by the learner and the educator. By keeping the experiences of the learner at the forefront, the opportunity is given to learn by doing and supported with feedback.

Preeclampsia is clinically defined as a blood pressure of 140/90 mmHg or above after the 20th week of pregnancy and the addition of proteinuria (300mg / 24 hours). It can develop in about 5-10% of all pregnancies. It is defined as a nulliparous disease since it is seen in approximately 85% of women during their first pregnancy. Preeclampsia constitutes 15% of the causes of maternal mortality in our country.

In studies evaluating the effectiveness of simulation training in planning the follow-up and care of preeclampsia, it was determined that this method increases the knowledge and self-confidence of nurses. For example; Christian and Krumwiede's study they found that the self-efficacy rates were significantly higher in the post-simulation test. In his study, Olubumno investigated the importance of simulation in increasing the critical thinking of perinatology nurses in the care of preeclamptic pregnant women, he found that the pre-test and post-test scores increased by 0.75 points, and this difference between the scores is statistically significant. Tabatabaeian et al., In their study comparing the effects of simulation-based education, coeducation and theoretical education on the performance of midwives in preeclampsia and eclampsia, found that the mean of the simulation group was higher than the other two groups.

Preeclampsia is an important obstetric emergency in women's health and disease nursing. Thus, when they start working in the clinic, it is aimed to be able to suspect preeclampsia with the anamnesis they received from the pregnant who applied to them, and to gain them with the simulation method what they should pay attention to and how to do in the follow-up of the pregnant woman hospitalized with the diagnosis of preeclampsia. Studies conducted in our country did not include studies involving students and healthcare professionals in the management of preeclampsia with simulation methods. Therefore, it is aimed to contribute to the literature with this study.

ELIGIBILITY:
Inclusion Criteria:

* Working for 1-5 years.
* Working in the gynecology inpatient services and delivery rooms of hospitals.
* To be a graduate nurse or midwife.
* Volunteering to participate in the study.

Exclusion Criteria:

* Being a high school graduate working in the related field
* Having just graduated from a related field

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-07-18 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
The level of knowledge about preeclamptic pregnancy care is higher in the group that received training with the lecturing and high-reality simulation method compared to the group that received training only with lectures | Six weeks
  "Self-efficacy for preeclamptic pregnancy care" scale was developed and used in the follow-up and care of preeclamptic pregnant women in order to evaluate the perception of self-efficacy towards nursing care in critical obstetric conditions related to preeclampsia in nurses and midwives. It's a 20-item instrument using a five-point scale.

SECONDARY OUTCOMES:
Educational Practices Questionnaire | One week after theoretical training
  The Educational Practices in Simulation Scale (EPSS), a 16-item instrument using a five-point scale, was designed to measure whether four educational practices (active learning, collaboration, diverse ways of learning, and high expectations) are present in the instructor-developed simulation, and the importance of each practice to the learner.
Student Satisfaction and Self-Confidence in Learning Scale | One week after theoretical training
  A total of 13 items assess the attitudes toward satisfaction with instruction and self-confidence in learning in simulation. A "satisfaction with instruction" subscale contains five items measuring satisfaction with teaching methods, diversity of learning materials, facilitation, motivation, and overall suitability of simulation. A "self-confidence with learning" subscale contains eight items measuring self-confidence in content mastery, content necessity, skills development, available resources, and knowledge of how to obtain help to solve clinical problems in simulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University Hospitals, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No